CLINICAL TRIAL: NCT04696679
Title: Quality of Life of Very Preterm Children With Dysexecutive Disorders at Elementary School Age During the Confinement-deconfinement Period of Covid-19 Pandemic
Acronym: GPE-QolVID
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-38; 2020-A01631-38 (Other: ANSM)
Record Dates: First submitted 2020-11-03; First posted 2021-01-06 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Very Preterm Children With Dysexecutive Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Very preterm children group
  Interventions: Other: Patient Quality of life assessment
- Control group
  Interventions: Other: Control group Quality of life assessment

INTERVENTIONS:
Other: Patient Quality of life assessment — Other: Patient questionnaire about quality of life assessment and their determinants during the confinement-deconfinement period of Covid-19 pandemic in France
  Groups: Very preterm children group
Other: Control group Quality of life assessment — Other: Patient questionnaire about quality of life assessment and their determinants during the confinement-deconfinement period of Covid-19 pandemic in France relationships with teachers, schoolwork, and self-esteem)
  Groups: Control group

SUMMARY:
Since March 2020, a new HCoV, SARS-Cov2, originating in China, has been spreading around the world. As of 13 may 2020, almost 4.2 million cases of infections and 292 000 died were reported worldwide (140 000 infection cases and 27 000 died in France). Human coronaviruses (HCoV) usually cause common upper respiratory tract infections in children and sometimes exacerbate lung and asthma diseases.

To minimize the risk of contamination of SARS-Cov2 (Covid-19), the French government has put in place directives that modified the daily lives of students, teachers and families. The societal change imposed by the state of health emergency with a confinement and deconfinement period could strongly impact the quality of life of very preterm children with dysexecutive disorders. These children are a population vulnerable to changes, especially during the pivotal period of elementary school. The executive dysfunctions disrupt children's learning and schooling, as well as their social adaptation, compromising their personal development and therefore, their quality of life.

ELIGIBILITY:
Very preterm children group :

* Children at elementary school age 7 to 9
* Children included in the cohort of EPIREMED study, born between 24 and 34 weeks' GA (gestational amenorrhea) and having visuospatial Working Memory impairment defined by a working memory index <85 from the WPPSI IV
* Children able to read, write and comprehend;
* Children whose parents are not opposed to the participation in the study
* Children affiliated to the French social security system

Control group :

* Children at elementary school age 7 to 9
* Children born at full-term and without dysexecutive disorders
* Children from the staff of the Assistance Publique - Hôpitaux de Marseille (AP-HM) / from the staff of the French Mediterranean network (PERINAT-MED) / from the close entourage of EPIREMED children
* Children able to read, write and comprehend
* Children whose parents are not opposed to the participation in the study
* Children affiliated to the French social security system

Ages: 7 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Children aged between 7 and 9
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the quality of life using the questionnaire Kidscreen 10 Index | 1 day
  The questionnaire Kidscreen 10 Index was developed in several European countries including France. It comprises 10 items from a version of 27 items, which explore the following domains: physical well-being, psychological well-being (positive and negative), autonomy and parents, peers and social support, and school environment
Assessment of the quality of life using The VSP-A questionnaire (Life and Perceived Health of the Adolescent and the Child) | 1 day
  The VSP-A questionnaire (Life and Perceived Health of the Adolescent and the Child) which groups together nine dimensions (vitality, psychological well-being, friendships, recreation, family relationships, physical well-being, relationships with teachers, schoolwork, and self-esteem)

SECONDARY OUTCOMES:
Specific data concerning the period of confinement-deconfinement | 1 day
  continuation of parental employment and current modalities: face-to-face, teleworking, part-time employment, etc.
  * possible schooling and current modalities: continued schooling, interruption of schooling, etc.
  * related ad hoc items to the state of health of the family unit, to medical events that have occurred (including family member(s) with a Covid-19 infection), to a history of hospitalization related to Covid-19 reasons, (reasons, consequences, frequency) between the beginning of the confinement and the moment they complete the questionnaire; as well as ad hoc items of anxiety related to Covid-19
Data on children behavioral disorders: | 1 day
  assessed by the Goodman questionnaire (Strengths and Difficulties Questionnaire)
Data concerning the anxiety symptoms of the parent completing the survey questionnaire: | 1 day
  assessed by the Spielberger questionnaire, as a personality trait and as an emotional state linked to the health protocol (State-Trait Anxiety Inventory, STAI)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique des Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided